CLINICAL TRIAL: NCT03531645
Title: A Pilot Phase II Study of Neoadjuvant Fulvestrant Plus Abemaciclib in Women With Advanced Low Grade Serous Carcinoma
Brief Title: Fulvestrant Plus Abemaciclib in Women With Advanced Low Grade Serous Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0405; NCI-2018-00941 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasms of Female Genital Organs
Keywords: Malignant neoplasms of female genital organs; Advanced low grade serous ovarian, primary peritoneal, or fallopian tube carcinomas; Fulvestrant; Faslodex; Abemaciclib; PD-0332991; Ibrance
MeSH Terms: interventions — Fulvestrant; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fulvestrant + Abemaciclib (Experimental)
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Fulvestrant — Neoadjuvant Treatment (Cycles 1-4): Fulvestrant 500 mg injection in buttocks on Days 1 and 15 of Cycle 1 and Day 1 of Cycles 2-4.
  Adjuvant Treatment (Cycles 5 and beyond): Fulvestrant 500 mg injection in buttocks on Day 1 of each cycle.
  Study cycle is 28 days.
  Other Names: Faslodex
Drug: Abemaciclib — Neoadjuvant Treatment (Cycles 1-4): Abemaciclib 150 mg by mouth On Days 1-28 of each cycle.
  Adjuvant Treatment (Cycles 5 and beyond): On Days 1-28 of each cycle, you will take Abemaciclib 150 mg by mouth on Days 1-28 of each cycle.
  Study cycle is 28 days.

SUMMARY:
The goal of this clinical research study is to learn if fulvestrant and abemaciclib can help to control low-grade serous ovarian cancer. The safety of this drug combination will also be studied.

This is an investigational study. Fulvestrant and abemaciclib are both FDA approved and commercially available for the treatment of several types of cancer. Their use in patients with low-grade serous ovarian cancer is investigational. The study doctor can explain how the study drugs are designed to work.

Up to 15 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration

Every study cycle will be 28 days. You will receive treatment in 2 periods: Neoadjuvant Treatment (before surgery) and Adjuvant Treatment (after surgery).

If you are premenopausal or perimenopausal, you will receive goserelin as an injection under the skin every 12 weeks. The study doctor will tell you if you will have these injections.

Neoadjuvant Treatment (Cycles 1-4) There are 4 cycles in the neoadjuvant treatment period. On Days 1 and 15 of Cycle 1 and Day 1 of Cycles 2-4, you will receive fulvestrant as an injection in your buttocks. On Days 1- 28 of each cycle, you will take abemaciclib tablets 2 times every day by mouth at about the same time each day, preferably with food.

Abemaciclib should be swallowed whole; not chewed. If a tablet is broken, cracked, or otherwise not whole, do not take it.

Surgery After 4 cycles of neoadjuvant treatment, you will have your scheduled surgery as part of your standard care. You will sign a separate consent for this surgery describing the procedure and its risks in more detail.

Adjuvant Treatment (Cycles 5 and beyond) After you have recovered from surgery (about 3-6 weeks later), you will begin receiving fulvestrant and abemaciclib. On Day 1 of each cycle, you will receive fulvestrant as an injection in your buttocks. On Days 1- 28 of each cycle, you will take abemaciclib tablets 2 times every day by mouth.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Length of Study You will receive the study drug(s) for as long as the study doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over after the 30-day follow-up phone call (described below).

Study Visits

On Day 1 of each cycle:

You will have a physical exam. If the study doctor thinks it is needed, you will also have a pelvic exam.

Blood (about 4 tablespoons) will be drawn for routine, tumor marker, and biomarker tests.

Urine will be collected for routine tests. If you can become pregnant, part of this blood sample will be used for a pregnancy test.

On Day 15 of Cycle 1, you will have a physical exam.

On Day 1 of odd-numbered cycles after Cycle 1 (Cycles 3, 5, 7, and so on), you will have an MRI or CT scan.

At your visit before the surgery, you will have a CT scan or MRI to check the status of the disease.

During surgery, some of the tissue removed will be used to compare to tissue collected from you before you received chemotherapy so researchers can learn if the study drugs had any affect on the disease. This sample will be stored at MD Anderson for an unlimited amount of time for testing related to this study.

End-of-Treatment Visit

After the last dose of study drug(s):

You will have a physical exam. Blood (about 1-2 tablespoons) will be drawn for routine, tumor marker, and biomarker tests.

You will have an MRI or CT scan to check the status of the disease.

Follow-Up About 30 days after the last dose of study drugs, the study staff will call you and ask how you are doing. This call should last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical or surgical stage III or IV low-grade serous ovarian, primary peritoneal, or fallopian tube carcinomas who in the judgement of the treating physician are unlikely to achieve optimal surgical cytoreduction and have been recommended to receive neoadjuvant therapy.
2. Histological diagnosis must be based on surgical or core biopsy not just fine needle aspiration. Biopsies performed at other institutions must undergo pathology review and confirmation at MD Anderson Cancer Center.
3. Tissue from an archival tissue sample or fresh tissue obtained from a core or excisional biopsy of a tumor lesion.
4. Willingness to provide pre- and post-treatment tissue for translational studies. Pre-treatment fresh frozen tissue must be available for research purposes. This tissue can be collected from preoperative laparoscopy, other diagnostic biopsy, or a research-specific biopsy.
5. Signed informed consent on protocol LAB02-188.
6. Tissue from an archival tissue sample or fresh tissue obtained from a core or excisional biopsy of a tumor lesion.
7. Patients whose clinical biopsies are found to be insufficient for the planned translational studies must be willing to undergo a research biopsy.
8. Patients must have measurable disease by RECIST v1.1. a. Measurable disease is defined at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each target lesion must be >20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or >10 mm when measured by spiral CT.
9. Women 18 years of age or older.
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
11. Abnormal organ function is permitted. However, patients must have: a. absolute neutrophil count >/= 1500/mL b. platelets >/= 100,000/mL c. hemoglobin >/= 9 g/dL d. estimated creatinine clearance >/= 60 ml/min as calculated using the method standard for the institution e. total serum bilirubin </= 1.5 X ULN f. aspartate aminotransferase (AST/SGOT) and/or alanine aminotransferase (ALT/SGPT) </= 3 X ULN (</= 5 X ULN in patients with bone or liver metastases)
12. Resolution of all acute toxic effects of prior therapy or surgical procedures to National Cancer Institute (NCI) CTCAE 4.03 Grade </= 1
13. Women of child-bearing potential (intact uterus) MUST have a negative serum or urine human chorionic gonadotropin (HCG) test within 72 hours prior to receiving the first dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 7.7). Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
15. Pre/perimenopausal women must be amenable to be treated with goserelin. All patients will be rendered post-menopausal secondary to concomitant administration of goserelin.
16. Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures.

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
3. Current use of food or drugs known to be potent CYP3A4 inhibitors, drugs known to be potent CYP3A4 inducers (for examples, see the Prohibited Concomitant Medications section), and drugs that are known to prolong the QT interval (see Prohibited Concomitant Medications in section 7.6.2).
4. Diagnosis of another malignancy within 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
5. Previous chemotherapy or hormonal therapy for treatment of ovarian cancer.
6. Known Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV) infection.
7. Inability or unwillingness to swallow pills.
8. Active infection requiring intravenous (IV) antibiotics or other uncontrolled intercurrent illness requiring hospitalization.
9. Inability to comply with the study and follow-up procedures.
10. History of any of the following: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), sudden cardiac arrest.
11. Prior hematopoietic stem cell or bone marrow transplantation.
12. Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding intramuscular injections of fulvestrant or goserelin (if applicable).
13. Known or possible hypersensitivity to fulvestrant, or abemaciclib or any of their excipients.
14. Pre/perimenopausal women with a known hypersensitivity to gnRH (gonadotropin-releasing hormone) agonists.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 112 days
  Clinical benefit rate determined by partial response (PR), complete response (CR), and stable disease (SD) associated with 4 cycles of neoadjuvant abemaciclib plus fulvestrant in patients with Low Grade Serous Carcinoma (LGSC). CBR assessed using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Amir A. Jazaeri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We are pending discussions with Eli Lilly and AstraZeneca regarding the level and quantity of data that may be shared. Discussions will also include potential modifications of the contract to allow for data sharing.

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org